CLINICAL TRIAL: NCT02280759
Title: Efficacy of Gelatin Tannate in Treatment Acute Gastroenteritis in Children: A Double Blind Randomized, Placebo- Controlled Trial .
Brief Title: Efficacy of Gelatin Tannate in Treatment Acute Gastroenteritis in Children.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KB56/2014
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Acute Gastroenteritis
Keywords: diarrhea, gelatin tannate, acute gastroenteritis
MeSH Terms: conditions — Diarrhea | interventions — tannate gelatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gelatin Tannate (Active Comparator): Gelatin Tannate:
  4 times 250 mg/daily for 5 days for children under 3. years old or 4 times 500mg/daily for 5 days for children older then 3. years and under 5 years.
  Interventions: Drug: Gelatin Tannate
- Placebo (Placebo Comparator): Placebo consists of an identical formulation, except active substance.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gelatin Tannate
  Arms: Gelatin Tannate
Drug: Placebo — Placebo consists of an identical formulation, except active substance
  Arms: Placebo

SUMMARY:
Gelatin tannate possesses astringent, antibacterial, and anti-inflammatory properties. It is increasingly being marketed as an antidiarrheal drug. A randomized, double blind, placebo-control trial was performed to assess the effectiveness of GT in management of children with acute gastroenteritis.

ELIGIBILITY:
Inclusion Criteria:

* children < 5 years old
* diarrhea (defined as the passage of 3 or more loose or watery stools per day) for > 1 day but < 5 days
* inform consent sign

Exclusion Criteria:

* regularly used antibiotics, probiotics, gelatin tannate, diosmectite, racecadotril within 7 days before admission
* underlying gastrointestinal tract disorder presenting with diarrhea
* breastfeeding >50%
* malnutrition (weight/high <3pc)

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-06-10 (Actual); Study Completion 2017-06-10 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea | 7 days
  time till the first normal stool from the onset of diarrhea or normalization number of stools and last those for 48hours

SECONDARY OUTCOMES:
Need of intravenous rehydration due to diarrhea | 7 days
Need of hospitalization in outpatients | 7 days
Vomiting | How many times for 7days
Weight gain | 7 days
Diarrhea recurrence | 7 days
Frequency of watery stools | 7 days
Adverse effects | 7 days
Severity of diarrhea due to modified Vesikari score | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Szajewska, Profesor, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Paediatrics, The Medical University of Warsaw, Poland, Warsaw, Poland

REFERENCES:
- [Derived] Kolodziej M, Bebenek D, Konarska Z, Szajewska H. Gelatine tannate in the management of acute gastroenteritis in children: a randomised controlled trial. BMJ Open. 2018 May 24;8(5):e020205. doi: 10.1136/bmjopen-2017-020205. PMID 29794092
- [Derived] Michalek D, Kolodziej M, Konarska Z, Szajewska H. Efficacy and safety of gelatine tannate for the treatment of acute gastroenteritis in children: protocol of a randomised controlled trial. BMJ Open. 2016 Feb 19;6(2):e010530. doi: 10.1136/bmjopen-2015-010530. PMID 26895988